CLINICAL TRIAL: NCT03592446
Title: Xidian University,China
Brief Title: Neural Alteration Response to Transcutaneous Auricular Vagus Nerve Stimulation (taVNS) in Depressed Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xidian University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 81471812
Record Dates: First submitted 2018-06-26; First posted 2018-07-19 (Actual); Last update posted 2018-07-19 (Actual); Status verified 2018-06

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active-raVNS (Experimental): Transcutaneous electrical vagus nerve stimulation at ear.
  Interventions: Device: Transcutaneous electrical vagus nerve stimulation
- Sham-raVNS (Sham Comparator): Sham vagus nerve stimulation at ear.
  Interventions: Device: Sham vagus nerve stimulation

INTERVENTIONS:
Device: Transcutaneous electrical vagus nerve stimulation — All subjects receive electrical VNS stimulation at cymba conchae.
  Arms: Active-raVNS
Device: Sham vagus nerve stimulation — All subjects receive electrical stimulation at earlobe.
  Arms: Sham-raVNS

SUMMARY:
Electrical vagus nerve stimulation (VNS) was approved by FDA for treatment of chronic recurrent depression in 2005. Recently, non-invasive, transcutaneous auricular vagus nerve stimulation （taVNS） has already been used for depression treatment. However, the neural mechanism remains unclear, and the relationship between stimulation parameters and neural response were also unknown. The present study aims to investigate the specific brain activation in depression patients after taVNS，compared with healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* Meets ICD-10 diagnosis standard;
* without taking anti-depressive medication or other psychiatric medications 2 weeks before the experiment;
* Patient has exhibited symptoms for at least 2 months, but no longer than 2 years.

Exclusion Criteria:

* With current addiction to drugs;
* With other severe organic diseases, such as severe heart disease, kidney failure etc;
* disagree with the consent form.
* Cannot receive MRI scan.

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2020-07-30 (Estimated); Study Completion 2020-07-30 (Estimated)

PRIMARY OUTCOMES:
actual neural activation in brain | 2 hours
  By using fMRI technology, the BOLD signal of brain is analyzed.

SECONDARY OUTCOMES:
Heart rate variability | 2 hours
  Frequency domain methods is used to analyze the bands of frequency and then count the number of NN intervals that match each band. The bands are typically high frequency (HF) from 0.15 to 0.4 Hz, low frequency (LF) from 0.04 to 0.15 Hz, and the very low frequency (VLF) from 0.0033 to 0.04 Hz.